CLINICAL TRIAL: NCT01102400
Title: A Phase I, Open-Label Study to Assess the Safety, Tolerability and Pharmacokinetics of Ascending Doses of MEDI-575 in Patients With Advanced Solid Malignancies
Brief Title: A Study of MEDI-575 in Patients With Advanced Solid Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D2840C00001
Record Dates: First submitted 2010-03-31; First posted 2010-04-13 (Estimated); Last update posted 2013-02-06 (Estimated); Status verified 2013-02

CONDITIONS: Advanced Solid Malignancies
Keywords: cancer; tumor; hepatocellular carcinoma
MeSH Terms: conditions — Neoplasms; Carcinoma, Hepatocellular | interventions — Tovetumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: MEDI-575

INTERVENTIONS:
Drug: MEDI-575 — MEDI-575 will be administered weekly or every 3 weeks as IV infusion as part of a 21-day treatment cycle. One or two doses will be selected for expansion part

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of MEDI-575 in Japanese patients with advanced solid tumors (dose escalation part) and hepatocellular carcinoma (expansion part).

ELIGIBILITY:
Inclusion Criteria:

* Having advanced solid malignancy for which no curative or standard therapies exist
* Karnofsky performance status of ≥60
* Patients must have histological confirmed diagnosis of HCC with no standard therapy available (for only expansion part)

Exclusion Criteria:

* Inadequate bone marrow reserve or organ function
* Major surgery within 4 weeks or minor surgery within 2 weeks prior to receipt of MEDI-575. Patients must have no unhealed wounds or unhealed fractures
* History of allergy or reaction to any component of the MEDI-575 and/or monoclonal antibody

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2010-03; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability assessed primarily by adverse events including abnormal values of clinical laboratory test, ECG and vital sign | 30 days after the last dose of MEDI-575

SECONDARY OUTCOMES:
Pharmacokinetic variables of MEDI-575 by assessment of drug concentrations in serum after intravenous infusion | 30 days after last dose of study drug
To evaluate the immunogenicity of MEDI-575 by measuring anti-MEDI-575 antibodies | 3 months after last dose of study drug
Anti-tumor activity of MEDI-575 using Response Evaluation Criteria in Solid Tumors (RECIST) | 3 months after last dose of study drug

CONTACTS AND LOCATIONS:
Locations (5):
- Japan (5):
  - Research Site, Nagoya, Aichi-ken
  - Research Site, Kashiwa, Chiba
  - Research Site, Matsuyama, Ehime
  - Research Site, Chuo-ku, Tokyo
  - Research Site, Sunto-gun

REFERENCES:
- [Derived] Murakami H, Ikeda M, Okusaka T, Inaba Y, Iguchi H, Yagawa K, Yamamoto N. A Phase I study of MEDI-575, a PDGFRalpha monoclonal antibody, in Japanese patients with advanced solid tumors. Cancer Chemother Pharmacol. 2015 Sep;76(3):631-9. doi: 10.1007/s00280-015-2832-6. Epub 2015 Jul 30. PMID 26223436